CLINICAL TRIAL: NCT04265157
Title: Hepato-duodenal Ligament Occlusion Versus Classic Technique During Recipient Hepatectomy in Liver Transplantation
Brief Title: Hepato-duodenal Ligament Occlusion and Classic Technique in Liver Transplant
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed mahmoud mohammed elkoussy, Assisstant lecturer, Assiut University
Other Study IDs: LDLT
Record Dates: First submitted 2020-01-29; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early occlusion of hepatoduodenal ligament: Early occlusion of hepatoduodenal ligament during mobilization of the liver of the recipient by using portal vein clamp or occlusive temporary bands.
  Interventions: Procedure: Surgical technique surgical occlusion
- classical occlusion of hepatoduodenal ligament: classical occlusion of hepatoduodenal ligament after mobilization of the liver of the recipient immediately before explantation by suing of portal vein clamp
  Interventions: Procedure: Surgical technique surgical occlusion

INTERVENTIONS:
Procedure: Surgical technique surgical occlusion — Occlusion of hepatoduodenal ligament by clamp or occlusive bands

SUMMARY:
Liver transplantation was historically associated with massive blood loss. Many factors have contributed to the decline in bleeding and transfusion in the past two decades including refinement of surgical techniques, anesthetics management and the use of point of care guided goal-directed hemostatic therapies. Increasing awareness of the adverse associations of allogenic transfusion has driven the quest for transfusion-free transplantation. Pre-operative management of preoperative anemia and targeted correction of coagulopathy is done to decrease blood transfusion. Liver transplantation is associated with the potential for massive operative blood loss, which has been recognized as one of the main causes of morbidity and mortality after liver transplantation. Therefore, a fine surgical procedure to reduce intraoperative hemorrhage is necessary for favorable outcomes of liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing Living Donor Liver Transplantation accepted according to hospital protocol
* All patients with liver Cirrhosis who have Porto systemic collaterals based on ct angiography

Exclusion Criteria:

* Acute fulminant liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will included in the study all patients accepted for Living Donor LiverTransplantation (LDLT) according to hospital protocol
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The amount of intraoperative blood loss measure by Cubic Cm | 2 hours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Donohue CI, Mallett SV. Reducing transfusion requirements in liver transplantation. World J Transplant. 2015 Dec 24;5(4):165-82. doi: 10.5500/wjt.v5.i4.165. PMID 26722645
- [Background] Park YK, Kim BW, Wang HJ, Xu W. Usefulness of the Pinch-Burn-Cut (PBC) technique for recipient hepatectomy in liver transplantation. Korean J Hepatobiliary Pancreat Surg. 2012 Feb;16(1):13-6. doi: 10.14701/kjhbps.2012.16.1.13. Epub 2012 Feb 29. PMID 26388900
- [Background] Houben P, Khajeh E, Hinz U, Knebel P, Diener MK, Mehrabi A. SEALIVE: the use of technical vessel-sealing devices for recipient hepatectomy in liver transplantation: study protocol for a randomized controlled trial. Trials. 2018 Jul 16;19(1):380. doi: 10.1186/s13063-018-2778-1. PMID 30012178
- [Background] Choi JU, Hwang S, Ahn CS, Moon DB, Ha TY, Kim KH, Song GW, Jung DH, Park GC, Lee SG. Prolonged occlusion of the hepatoduodenal ligament to reduce risk of bleeding and tumor spread during recipient hepatectomy for living donor liver transplantation. Ann Hepatobiliary Pancreat Surg. 2019 Feb;23(1):61-64. doi: 10.14701/ahbps.2019.23.1.61. Epub 2019 Feb 28. PMID 30863809
- [Background] Lee KF, Wong J, Cheung SYS, Chong CCN, Hui JWY, Leung VYF, Yu SCH, Lai PBS. Does Intermittent Pringle Maneuver Increase Postoperative Complications After Hepatectomy for Hepatocellular Carcinoma? A Randomized Controlled Trial. World J Surg. 2018 Oct;42(10):3302-3311. doi: 10.1007/s00268-018-4637-3. PMID 29696328
- [Background] Cleland S, Corredor C, Ye JJ, Srinivas C, McCluskey SA. Massive haemorrhage in liver transplantation: Consequences, prediction and management. World J Transplant. 2016 Jun 24;6(2):291-305. doi: 10.5500/wjt.v6.i2.291. PMID 27358774
- [Background] Yoon JU, Byeon GJ, Park JY, Yoon SH, Ryu JH, Ri HS. Bloodless living donor liver transplantation: Risk factors, outcomes, and diagnostic predictors. Medicine (Baltimore). 2018 Dec;97(50):e13581. doi: 10.1097/MD.0000000000013581. PMID 30558025
- [Background] Kornberg A, Witt U, Kornberg J, Ceyhan GO, Mueller K, Friess H, Thrum K. Prognostic Impact of Intraoperative Blood Loss in Liver Transplant Patients with Advanced Hepatocellular Carcinoma. Anticancer Res. 2016 Oct;36(10):5355-5364. doi: 10.21873/anticanres.11109. Epub 2016 Oct 10. PMID 27798899